CLINICAL TRIAL: NCT03480594
Title: Effect of Fatty Liver on TCA Cycle Flux and the Pentose Phosphate Pathway (HP FFF)
Brief Title: Effect of Fatty Liver on TCA Cycle Flux and the Pentose Phosphate Pathway
Acronym: HPFFF
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Principal Investigator, Craig Riggs Malloy, Principal Investigator, University of Texas Southwestern Medical Center
Other Study IDs: 082017-019; 5P41EB015908-30 (NIH)
Record Dates: First submitted 2018-03-21; First posted 2018-03-29 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Fatty Liver
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Fatty Liver Patients: Hyperpolarized [13C] Pyruvate Injection in Fatty Liver patients
  Interventions: Drug: MRI Tracer
- Healthy Control Subjects: Hyperpolarized [13C] Pyruvate Injection in Healthy Control Subjects
  Interventions: Drug: MRI Tracer

INTERVENTIONS:
Drug: MRI Tracer — Hyperpolarized [1-13C] pyruvate for injection under IND133229 used to enhance MRI/MRS/MRSI using a 3T MRI scanner.

SUMMARY:
The investigators plan to evaluate sensitivity and specificity of HP 13C-pyruvate as an imaging agent for detection of altered PDH flux in fatty liver.

DETAILED DESCRIPTION:
The investigators plan to determine whether nutritional state and fatty liver influence the production of [13C]bicarbonate from [1-13C]pyruvate via flux through the pyruvate dehydrogenase (PDH) reaction in healthy subjects compared to those with fatty liver. The long-term purpose of this work is to develop hyperpolarized 13C imaging as a method to directly assess metabolic pathways in the human liver. Many high-impact diseases such as insulin resistant states, fatty liver and inborn errors of metabolism are known to alter biochemical fluxes and for this reason it is important to detect altered activity in specific pathways.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 99 years.
* All races, ethnicities and gender identification may be included. Subjects must meet all of the inclusion and exclusion criteria to be included in the study.
* Either fatty liver diagnosis (defined as >5.6% fat content in the liver) or healthy control
* While all races and ethnicities will be included, subjects must be able to read and speak the English language. Once the protocol is established, Spanish-speaking participants will be included.
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Exclusion Criteria:

Fatty Liver Subjects

* No subjects taking hypoglycemic agents or insulin will be enrolled. There is no exclusion based on fasting glucose.
* Subjects with major mental health conditions such as schizophrenia and bipolar disorder that would limit compliance with study requirements will not participate. In general, subjects with any form of medical instability such as seizure disorders, significant COPD, significant asthma, left ventricular dysfunction will not participate.
* Medications for control of hypercholesterolemia, hypertriglyceridemia or hyperglycemia.

Healthy Control Subjects

* Liver disease or other chronic illness
* Diagnosis of type I or type II diabetes
* No subjects taking hypoglycemic agents or insulin will be enrolled. There is no exclusion based on fasting glucose.
* A potential subject with any major medical, surgical or psychiatric condition will not participate. These conditions include but are not limited to thyroid disease, chronic metabolic illness, known vascular disease, current cancer diagnosis and/or treatment.
* Subjects with major mental health conditions such as schizophrenia and bipolar disorder that would limit compliance with study requirements will not participate. In general, subjects with any form of medical instability such as seizure disorders, significant COPD, significant asthma, left ventricular dysfunction will not participate.
* Medications for control of hypercholesterolemia, hypertriglyceridemia or hyperglycemia.

All Subjects

* No prior hepato-biliary surgery.
* Donated blood within the prior 4 weeks.
* Consume more than 10 grams of ethanol per day.
* Cirrhosis or any form of viral hepatitis.
* Prior documented hepatic reaction to drugs with a known hepatotoxicity profile such as isoniazid, methotrexate, phenytoin, propylthiouracil, valproate, etc.
* Pregnant/Lactating
* Receiving any other investigational agents.
* Any contraindication noted on the UTSWMC MRI Screening Form including implants contraindicated at 3T, pacemakers, Implantable Cardioverter Defibrillators (ICD), etc., and significant claustrophobia.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The plan is to study fatty liver patients and healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
Bicarbonate:lactate ratio | One visit of 6 hours; two injections of HP pyruvate with MRI over 3 hours
  1. The ratio of hyperpolarized [13C]bicarbonate relative to hyperpolarized [1-13C]lactate. This measurement will be monitored from the subject's liver over a ~4 minute period in the MRI system.

SECONDARY OUTCOMES:
Labeled glycerol fraction | One visit of 6 hours; ingestion of Oral Glycerol with blood draws over 3 hours
  2. The fraction of [U-13C]glycerol that has passed through mitochondrial pathways prior to gluconeogenesis and the fraction of glucose, derived from [U-13C]glycerol, that has passed through the pentose phosphate pathway. This information will be acquired from 13C NMR spectroscopy of glucose and triglycerides from a venous blood sample, obtained after the hyperpolarization exam.

CONTACTS AND LOCATIONS:
Locations (1):
- Advanced Imaging Research Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ardenkjaer-Larsen JH, Fridlund B, Gram A, Hansson G, Hansson L, Lerche MH, Servin R, Thaning M, Golman K. Increase in signal-to-noise ratio of > 10,000 times in liquid-state NMR. Proc Natl Acad Sci U S A. 2003 Sep 2;100(18):10158-63. doi: 10.1073/pnas.1733835100. Epub 2003 Aug 20. PMID 12930897
- [Background] Nelson SJ, Kurhanewicz J, Vigneron DB, Larson PE, Harzstark AL, Ferrone M, van Criekinge M, Chang JW, Bok R, Park I, Reed G, Carvajal L, Small EJ, Munster P, Weinberg VK, Ardenkjaer-Larsen JH, Chen AP, Hurd RE, Odegardstuen LI, Robb FJ, Tropp J, Murray JA. Metabolic imaging of patients with prostate cancer using hyperpolarized [1-(1)(3)C]pyruvate. Sci Transl Med. 2013 Aug 14;5(198):198ra108. doi: 10.1126/scitranslmed.3006070. PMID 23946197
- [Background] Cunningham CH, Lau JY, Chen AP, Geraghty BJ, Perks WJ, Roifman I, Wright GA, Connelly KA. Hyperpolarized 13C Metabolic MRI of the Human Heart: Initial Experience. Circ Res. 2016 Nov 11;119(11):1177-1182. doi: 10.1161/CIRCRESAHA.116.309769. Epub 2016 Sep 15. PMID 27635086
- [Background] Neeland IJ, Hughes C, Ayers CR, Malloy CR, Jin ES. Effects of visceral adiposity on glycerol pathways in gluconeogenesis. Metabolism. 2017 Feb;67:80-89. doi: 10.1016/j.metabol.2016.11.008. Epub 2016 Nov 27. PMID 28081781
- [Background] Neuschwander-Tetri BA, Caldwell SH. Nonalcoholic steatohepatitis: summary of an AASLD Single Topic Conference. Hepatology. 2003 May;37(5):1202-19. doi: 10.1053/jhep.2003.50193. PMID 12717402
- [Background] Satapati S, Kucejova B, Duarte JA, Fletcher JA, Reynolds L, Sunny NE, He T, Nair LA, Livingston KA, Fu X, Merritt ME, Sherry AD, Malloy CR, Shelton JM, Lambert J, Parks EJ, Corbin I, Magnuson MA, Browning JD, Burgess SC. Mitochondrial metabolism mediates oxidative stress and inflammation in fatty liver. J Clin Invest. 2015 Dec;125(12):4447-62. doi: 10.1172/JCI82204. Epub 2015 Nov 16. PMID 26571396
- [Background] Satapati S, Sunny NE, Kucejova B, Fu X, He TT, Mendez-Lucas A, Shelton JM, Perales JC, Browning JD, Burgess SC. Elevated TCA cycle function in the pathology of diet-induced hepatic insulin resistance and fatty liver. J Lipid Res. 2012 Jun;53(6):1080-92. doi: 10.1194/jlr.M023382. Epub 2012 Apr 9. PMID 22493093
- [Background] Sunny NE, Parks EJ, Browning JD, Burgess SC. Excessive hepatic mitochondrial TCA cycle and gluconeogenesis in humans with nonalcoholic fatty liver disease. Cell Metab. 2011 Dec 7;14(6):804-10. doi: 10.1016/j.cmet.2011.11.004. PMID 22152305
- [Background] Jones JG. Hepatic glucose and lipid metabolism. Diabetologia. 2016 Jun;59(6):1098-103. doi: 10.1007/s00125-016-3940-5. Epub 2016 Apr 5. PMID 27048250
- [Background] Jin ES, Moreno KX, Wang JX, Fidelino L, Merritt ME, Sherry AD, Malloy CR. Metabolism of hyperpolarized [1-(13)C]pyruvate through alternate pathways in rat liver. NMR Biomed. 2016 Apr;29(4):466-74. doi: 10.1002/nbm.3479. Epub 2016 Feb 2. PMID 26836042
- [Background] Jin ES, Sherry AD, Malloy CR. An Oral Load of [13C3]Glycerol and Blood NMR Analysis Detect Fatty Acid Esterification, Pentose Phosphate Pathway, and Glycerol Metabolism through the Tricarboxylic Acid Cycle in Human Liver. J Biol Chem. 2016 Sep 2;291(36):19031-41. doi: 10.1074/jbc.M116.742262. Epub 2016 Jul 18. PMID 27432878
- [Background] Jin ES, Sherry AD, Malloy CR. Interaction between the pentose phosphate pathway and gluconeogenesis from glycerol in the liver. J Biol Chem. 2014 Nov 21;289(47):32593-603. doi: 10.1074/jbc.M114.577692. Epub 2014 Oct 6. PMID 25288790
- [Background] Lee P, Leong W, Tan T, Lim M, Han W, Radda GK. In vivo hyperpolarized carbon-13 magnetic resonance spectroscopy reveals increased pyruvate carboxylase flux in an insulin-resistant mouse model. Hepatology. 2013 Feb;57(2):515-24. doi: 10.1002/hep.26028. Epub 2013 Jan 10. PMID 22911492
- [Background] Moreno KX, Moore CL, Burgess SC, Sherry AD, Malloy CR, Merritt ME. Production of hyperpolarized 13CO2 from [1-13C]pyruvate in perfused liver does reflect total anaplerosis but is not a reliable biomarker of glucose production. Metabolomics. 2015 Oct;11(5):1144-1156. doi: 10.1007/s11306-014-0768-1. Epub 2015 Jan 9. PMID 26543443
- [Background] Merritt ME, Harrison C, Sherry AD, Malloy CR, Burgess SC. Flux through hepatic pyruvate carboxylase and phosphoenolpyruvate carboxykinase detected by hyperpolarized 13C magnetic resonance. Proc Natl Acad Sci U S A. 2011 Nov 22;108(47):19084-9. doi: 10.1073/pnas.1111247108. Epub 2011 Nov 7. PMID 22065779
- [Background] Moreno KX, Satapati S, DeBerardinis RJ, Burgess SC, Malloy CR, Merritt ME. Real-time detection of hepatic gluconeogenic and glycogenolytic states using hyperpolarized [2-13C]dihydroxyacetone. J Biol Chem. 2014 Dec 26;289(52):35859-67. doi: 10.1074/jbc.M114.613265. Epub 2014 Oct 28. PMID 25352600
- [Background] Moreno KX, Harrison CE, Merritt ME, Kovacs Z, Malloy CR, Sherry AD. Hyperpolarized delta-[1-13 C]gluconolactone as a probe of the pentose phosphate pathway. NMR Biomed. 2017 Jun;30(6):10.1002/nbm.3713. doi: 10.1002/nbm.3713. Epub 2017 Mar 8. PMID 28272754
- [Background] Jin ES, Szuszkiewicz-Garcia M, Browning JD, Baxter JD, Abate N, Malloy CR. Influence of liver triglycerides on suppression of glucose production by insulin in men. J Clin Endocrinol Metab. 2015 Jan;100(1):235-43. doi: 10.1210/jc.2014-2404. PMID 25250633
- [Background] Hensley CT, Faubert B, Yuan Q, Lev-Cohain N, Jin E, Kim J, Jiang L, Ko B, Skelton R, Loudat L, Wodzak M, Klimko C, McMillan E, Butt Y, Ni M, Oliver D, Torrealba J, Malloy CR, Kernstine K, Lenkinski RE, DeBerardinis RJ. Metabolic Heterogeneity in Human Lung Tumors. Cell. 2016 Feb 11;164(4):681-94. doi: 10.1016/j.cell.2015.12.034. Epub 2016 Feb 4. PMID 26853473
- [Background] Pichumani K, Mashimo T, Vemireddy V, Kovacs Z, Ratnakar J, Mickey B, Malloy CR, DeBerardinis RJ, Bachoo RM, Maher EA. Hepatic gluconeogenesis influences (13)C enrichment in lactate in human brain tumors during metabolism of [1,2-(13)C]acetate. Neurochem Int. 2016 Jul;97:133-6. doi: 10.1016/j.neuint.2016.03.015. Epub 2016 Mar 26. PMID 27020407
- [Background] Cheshkov S, Dimitrov IE, Jakkamsetti V, Good L, Kelly D, Rajasekaran K, DeBerardinis RJ, Pascual JM, Sherry AD, Malloy CR. Oxidation of [U-13 C]glucose in the human brain at 7T under steady state conditions. Magn Reson Med. 2017 Dec;78(6):2065-2071. doi: 10.1002/mrm.26603. Epub 2017 Jan 23. PMID 28112825